CLINICAL TRIAL: NCT02453854
Title: Study Protocol: Small Changes, a One-year Weight Management Intervention for Adults Who Are Overweight or Obese
Brief Title: Small Changes a One Year Protocol for Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Small Changes (Other)
Responsible Party: Principal Investigator, Trevor Simper, Dr Trevor Simper, Small Changes
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: smallchanges2011
Record Dates: First submitted 2015-05-18; First posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as Usual (Active Comparator): A Treatment as Usual (TAU) group received a psycho-educational programme for weight management over one year
  Interventions: Behavioral: Group motivational interviewing
- Group Motivational Intervieiwng (Experimental): A Motivational interviewing group received one year of programme using motivational interviewing as the approach for treatment.
  Interventions: Behavioral: Group motivational interviewing

INTERVENTIONS:
Behavioral: Group motivational interviewing — Monthly group meetings were held for two hour sessions each month and verifiable (treatment fidelity checked) motivational interviewing employed in helping clients make health behaviour changes.

SUMMARY:
A trial comparing Treatment as usual with Motivational Interviewing focussed treatment in the 'Small Changes' programme.

DETAILED DESCRIPTION:
A quasi-experimental design. With one arm focussed on 'treatment as usual' and the other on Motivational Interviewing. Subjects were not randomly assigned but treated as two separate cohorts one Running October 2011-October 2012 using the Treatment as usual and a separate cohort running from October 2012 to October -2013 using motivational interviewing as the approach for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass index equal to or greater than 30 kgm2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
weight | 1 year
  Bodyweight in Kilograms